CLINICAL TRIAL: NCT02700555
Title: Surveillance of Metabolic Parameters in Patients Who Will Receive Chemotherapy After Surgical Resection of Colorectal Cancer: KBSMC Colon Cancer Cohort
Brief Title: Surveillance of Metabolic Parameters in Patients With Colorectal Cancer
Acronym: SPRING
Status: Terminated | Type: Observational
Why Stopped: The patient's study enrollment was too low.
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Dong-Hoe Koo, Assistant Professor, Kangbuk Samsung Hospital
Other Study IDs: SPRING
Record Dates: First submitted 2016-02-24; First posted 2016-03-07 (Estimated); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; diabetes; metabolic parameters; Surveillance
MeSH Terms: conditions — Colorectal Neoplasms; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Biospecimen Retention: Samples Without DNA — Tumor tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
A prospective, single center, cohort study for surveillance of metabolic parameters in patients who will receive chemotherapy after surgical resection of colorectal cancer

DETAILED DESCRIPTION:
Primary objective - Incidence of newly developed diabetes mellitus in patients with colorectal cancer after post-operative chemotherapy

Secondary objective - Pre-operative incidence of diabetes and characteristics of metabolic parameters of patients with colorectal cancer; Incidence of developed poorly controlled glucose level in diabetic patients with colorectal cancer after post-operative chemotherapy; 3-year recurrence-free survival according to status of diabetes and metabolic parameters; 5-year recurrence-free survival according to status of diabetes and metabolic parameters

ELIGIBILITY:
Inclusion Criteria:

* Who will get surgical resection for colorectal cancer
* Who has diagnosed with diabetes
* Who met the criteria for testing of diabetes in asymptomatic adult individuals
* Criteria for testing for diabetes in asymptomatic adult individuals

  * overweight (BMI>25 kg/m2*) and have additional risk factors (physical inactivity, first-degree relative with diabetes, high-risk race/ethnicity (e.g., African American, Latino, Native American, Asian American, Pacific Islander), women who delivered a baby weighing 0.9 lb or were diagnosed with GDM, hypertension (>140/90 mmHg or on therapy for hypertension), HDL cholesterol level ,35 mg/dL (0.90 mmol/L) and/or a triglyceride level >250 mg/dL (2.82 mmol/L), women with polycystic ovarian syndrome, HbA1C >5.7%, IGT, or IFG on previous testing, other clinical conditions associated with insulin resistance (e.g., severe obesity, acanthosis nigricans), history of CVD)

Exclusion Criteria:

* Previously exposed to surgery or chemotherapy for colorectal cancer
* Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or prior malignancy treated more than 5 years ago without recurrence
* Presence of CNS metastasis
* Not able or willing to give informed consent
* Any patients judged by the investigator to be unfit to participate in the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will receive chemotherapy after surgical resection of colorectal cancer
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Incidence of newly developed diabetes mellitus | up to 12 months
  Incidence of newly developed diabetes mellitus in patients with colorectal cancer after post-operative chemotherapy

SECONDARY OUTCOMES:
Pre-operative incidence of diabetes | up to 12 months
  Pre-operative incidence of diabetes (> 6.5% of HbA1c) and abnormal metabolic parameters (> 23 kg/m2 of BMI or dyslipidemia) of patients with colorectal cancer;
Incidence of developed poorly controlled glucose level | up to 12 months
  Incidence of developed poorly controlled glucose level in diabetic patients with colorectal cancer after post-operative chemotherapy;
3-year recurrence-free survival & 5-year recurrence-free survival | up to 36-60 months
  3-year and 5-year recurrence-free survival according to status of diabetes (> 6.5% of HbA1c) and abnormal metabolic parameters (> 23 kg/m2 of BMI or dyslipidemia)

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Hoe Koo, MD,PhD, Principal Investigator — Kangbuk Samsung Hospital, Sungkyunkwan University School of Medicine
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Haggar FA, Boushey RP. Colorectal cancer epidemiology: incidence, mortality, survival, and risk factors. Clin Colon Rectal Surg. 2009 Nov;22(4):191-7. doi: 10.1055/s-0029-1242458. PMID 21037809
- [Background] Meyerhardt JA, Catalano PJ, Haller DG, Mayer RJ, Macdonald JS, Benson AB 3rd, Fuchs CS. Impact of diabetes mellitus on outcomes in patients with colon cancer. J Clin Oncol. 2003 Feb 1;21(3):433-40. doi: 10.1200/JCO.2003.07.125. PMID 12560431
- [Background] Mills KT, Bellows CF, Hoffman AE, Kelly TN, Gagliardi G. Diabetes mellitus and colorectal cancer prognosis: a meta-analysis. Dis Colon Rectum. 2013 Nov;56(11):1304-19. doi: 10.1097/DCR.0b013e3182a479f9. PMID 24105007
- [Background] Dienstmann R, Salazar R, Tabernero J. Personalizing colon cancer adjuvant therapy: selecting optimal treatments for individual patients. J Clin Oncol. 2015 Jun 1;33(16):1787-96. doi: 10.1200/JCO.2014.60.0213. Epub 2015 Apr 27. PMID 25918287
- [Background] Hwang JL, Weiss RE. Steroid-induced diabetes: a clinical and molecular approach to understanding and treatment. Diabetes Metab Res Rev. 2014 Feb;30(2):96-102. doi: 10.1002/dmrr.2486. PMID 24123849
- [Background] Feng JP, Yuan XL, Li M, Fang J, Xie T, Zhou Y, Zhu YM, Luo M, Lin M, Ye DW. Secondary diabetes associated with 5-fluorouracil-based chemotherapy regimens in non-diabetic patients with colorectal cancer: results from a single-centre cohort study. Colorectal Dis. 2013 Jan;15(1):27-33. doi: 10.1111/j.1463-1318.2012.03097.x. PMID 22594556
- [Background] American Diabetes Association. Standards of medical care in diabetes--2014. Diabetes Care. 2014 Jan;37 Suppl 1:S14-80. doi: 10.2337/dc14-S014. No abstract available. PMID 24357209